CLINICAL TRIAL: NCT02574130
Title: Effect of Additional Nebulized Amikacin in Ventilator-Associated Pneumonia Caused by Gram Negative Bacteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Pitchayapa Ruchiwit, Principal investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTU-EC-IM-2-046/57
Record Dates: First submitted 2015-10-09; First posted 2015-10-12 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Amikacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nebulized amikacin (Experimental): Amikacin 400 mg nebulized every 12 hours plus intravenous antibiotic(s) for 10 days
  Interventions: Drug: Amikacin
- placebo (Placebo Comparator): nebulized placebo every 12 hours plus intravenous antibiotic(s)for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amikacin — 400 mg, nebulizer, every 12 hours, 10 days
  Other Names: Amikin
  Arms: Nebulized amikacin
Drug: Placebo — placebo 4 ml, nebulizer, every 12 hours, 10 days
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the cure rate from ventilator-associated pneumonia (VAP) caused by Gram negative bacteria when administering add on nebulized amikacin to intravenous antibiotics compared to intravenous antibiotics alone.

DETAILED DESCRIPTION:
After inclusion, the patients are randomized into two groups: nebulized amikacin plus intravenous antibiotic(s) or nebulized placebo plus intravenous antibiotic(s). The dose of nebulized amikacin is 400 mg every 12 hours for 10 days. The patients are followed up on day 3, 7, 10, and 28 for safety and efficacy. The estimate sample size is 84 subjects base on previous study of cure rate in VAP and the authors expected that nebulized amikacin can improve cure rate in VAP subjects for 30% when compared with intravenous antibiotic(s) alone with power of 80% at level of significance 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* On mechanical ventilator more than 7 days
* VAP diagnosis inclusion criteria:

  1. new/progressive infiltration of chest radiography
  2. 2/3 of the following: 1) fever 2) purulent sputum 3) Wbc > 12,000 cell/mm3 or < 4,000 cell/mm3
* Evidence of gram negative bacilli from sputum gram stain or previous sputum culture within 1 week

Exclusion Criteria:

* History of amikacin allergy
* GFR < 30 mL/min except dialytic patients
* Immunocompromised host: HIV CD4 < 200 cells/mm3, leukemia, lymphoma, received chemotherapy within 3 weeks, Absolute neutrophil count < 500/mm3
* Severe ARDS (P/F ratio < 100)
* Endobronchial obstruction:endobronchial mass, endobronchial stenosis
* Atelectasis
* Severe bronchospasm
* Lung abscess
* Complicated parapneumonic effusion/ Empyema
* Chest trauma
* Uncontrolled extrapulmonary infection(s)
* Received intravenous antibiotic(s) more than 48 hours
* Pregnancy/ Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
cure rate | 10 days after end of the intervention
  Cure rate = improvement/ no new infiltration of chest radiography plus 2/3 of the following: 1) No fever within 48 hours after end of the intervention 2) The reduction of secretion 3) The reduction of white blood cell

SECONDARY OUTCOMES:
The reduction of pathogens | 10 days after end of the intervention
  quantitative sputum cultures were measured every days for 10 days or no growth of organism.
mortality rate | at 28 days after end of the intervention
  All causes of death during the intervention
duration of mechanical ventilation | at 28 days after end of the intervention
  number of days on mechanical ventilation
duration of ICU stay | at 28 days after end of the intervention
  number of ICU days
duration of hospitalization | at 28 days after end of the intervention
  number of days hospitalization
Safety of intervention drug | at 28 days after end of the intervention
  Any adverse events were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Pitchayapa Ruchiwit, MD, Principal Investigator — Thammasat University Hospital
Locations (1):
- Thammasat University (Rangsit center), Pathum Thani, Thailand

REFERENCES:
- [Result] Czosnowski QA, Wood GC, Magnotti LJ, Croce MA, Swanson JM, Boucher BA, Fabian TC. Adjunctive aerosolized antibiotics for treatment of ventilator-associated pneumonia. Pharmacotherapy. 2009 Sep;29(9):1054-60. doi: 10.1592/phco.29.9.1054. PMID 19698010
- [Result] Ghannam DE, Rodriguez GH, Raad II, Safdar A. Inhaled aminoglycosides in cancer patients with ventilator-associated Gram-negative bacterial pneumonia: safety and feasibility in the era of escalating drug resistance. Eur J Clin Microbiol Infect Dis. 2009 Mar;28(3):253-9. doi: 10.1007/s10096-008-0620-5. Epub 2008 Aug 28. PMID 18752007
- See also: Adjunctive aerosolized antibiotics for treatment of ventilator-associated pneumonia — https://www.ncbi.nlm.nih.gov/pubmed/19698010
- See also: Inhaled aminoglycosides in cancer patients with ventilator-associated Gram-negative bacterial pneumonia: safety and feasibility in the era of escalating drug resistance — https://www.ncbi.nlm.nih.gov/pubmed?term=Eur.+J.+Clin.+Microbiol.+Infect.+Dis%5BJour%5D+AND+Ghannam+DE%5Bauthor%5D&cmd=detailssearch